CLINICAL TRIAL: NCT03137251
Title: Evaluation of the Effectiveness of Transcutaneous Electrical Nerve Stimulation During Labor. A Triple Blind Randomized Clinical Trial
Brief Title: Evaluation of the Effectiveness of Transcutaneous Electrical Nerve Stimulation During Labor.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Las Palmas de Gran Canaria (Other)
Responsible Party: Principal Investigator, Aníbal Báez Suárez, Physiotherapist, University of Las Palmas de Gran Canaria
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ABSuarez
Record Dates: First submitted 2017-04-22; First posted 2017-05-02 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Midwifery; Pregnancy
Keywords: Transcutaneous electrical nerve stimulation; TENS; Analgesia; Labour pain; Physical therapy modality
MeSH Terms: conditions — Agnosia; Labor Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TENS 1 (Experimental): This group will receive TENS continuously for 30 minutes starting at the beginning of the active phase of labour.
  Dose TENS 1: Biphasic asymmetric pulse, pulse width of 100 µs and a frequency of 100 Hz. The intensity is individually titrated according to the sensitivity of the parturient.
  Interventions: Device: TENS 1; Device: TENS 2
- TENS 2 (Experimental): This group will receive TENS continuously for 30 minutes starting at the beginning of the active phase of labour.
  Dose TENS 2: Biphasic asymmetric pulse, pulse width of 350 µs and a variable frequency between 80 and 100Hz. The intensity is individually titrated according to the sensitivity of the parturient.
  Interventions: Device: TENS 2; Device: Placebo TENS
- Placebo TENS (Sham Comparator): This group will receive TENS continuously for 30 minutes starting at the beginning of the active phase of labour. However, TENS has been modified, so that it emits light and sound but does not transmit electrical current.
  Interventions: Device: TENS 1; Device: Placebo TENS

INTERVENTIONS:
Device: TENS 1 — A portable TENS unit will be used by the principal investigator to apply the experimental intervention. Two pairs of electrodes measuring 5 x 9 cm will be fixed on the paravertebral regions of the participants of the experimental group using hypoallergenic surgical tape. Two paired electrodes will be placed 1 cm laterally on either side of the spine at the T10 to L1 and S2 to S4 levels.
  Arms: Placebo TENS; TENS 1
Device: TENS 2 — An intervention similar to arm 1 will be performed but with different doses.
  Arms: TENS 1; TENS 2
Device: Placebo TENS — An intervention similar to arm 1and 2 will be performed but,in this case, it is a sham device.
  Arms: Placebo TENS; TENS 2

SUMMARY:
This study evaluates the effectiveness of the Transcutaneus Electric Nerve Stimulation (TENS) during the labour. TENS is a low frequency electrotherapy technique, analgesic type, generally used in musculoskeletal pathology.

The investigators will have three groups of participants to be administered the TENS, a different dose in two groups, while the third will correspond to placebo.

The hypothesis of the study is to verify if the TENS is effective as a non-pharmacological method in the relief of pain during childbirth

DETAILED DESCRIPTION:
1. Background:

   Pain during labour is one of the most intense pain that many women could experience during their lives, and it can be influenced by the anatomical and physiological factors of the labouring women, and also, by their psychological experiences, as well as by cultural, social, and environmental factors.

   Neuraxial analgesia during labour is the most effective method for pain relief, but it appears to be associated with certain side effects, such as maternal hypotension, decreased uteroplacental perfusion, foetal bradycardia, fever, pruritus, an increased oxytocin requirement, a prolonged second stage of labour, a higher rate of operative delivery, and high costs.

   The use of non-pharmacological methods for pain relief includes a wide variety of techniques aimed at improving physical sensations and preventing psychoemotional perception of pain. Among the main nonpharmacological methods of pain relief at delivery is the application of Transcutaneous electrical nerve stimulation (TENS). Its application during childbirth is based on the Gait Control theory of pain of Melzack and Wall. According to their theory, the application of TENS reduces the excitability of the delta A and C pain fibers, thus reducing the amount of painful messages ascending the spinal cord. Activation of these fibers stimulates the release of natural pain inhibitors.

   Furthermore, many non-pharmacological methods of managing pain increase the satisfaction of women with their childbirth experience.

   TENS have used for labour analgesia and there are several studies which show its effectiveness. The effectiveness of TENS depends on the duration, frequency and amplitude of the stimulating current and the site of application of the electrodes. TENS can be administered by either dermatomal stimulation or by stimulation of acupuncture points for labour analgesia. In addition, all studies stated that it was safe and there was no side effects on the mother and the baby.

   This work was conducted to study the effectiveness of TENS on labour analgesia, maternal and fetal outcome using TENS by dermatomal stimulation technique. Thus, device will be used as follows:

   Through electrodes applied to the lower back, the parturient can control both parameters, the frequency and intensity of the low-voltage electrical impulses emitted from the TENS device. When applying to the lower back, the TENS unit emits electrical impulses which excite afferent nerves, and thus inhibit the transmission of painful stimuli arising from the uterus, vagina and perineum during labour. These electrodes are attached to the skin bilaterally at paravertebral positions T10 and S2.

   In the present study the investigators will use three equal devices (two different dose and one placebo) .They will be assigned a number that associate to each group of participants.

   Safety profile in the use of TENS:

   It is a non-invasive technique, easy to administer, without side effects or interactions with other drugs, it cannot produce toxicity in the tissue or cellular level.

   The current literature does not reflect any complications, either on the part of the pregnant woman and in the fetus, during the application of TENS in the labor phase.

   The use of TENS should be contraindicated in women whose gestational age does not exceed 37 weeks, women with pacemakers and water births. It should not be applied in the maternal abdomen, at any time during pregnancy or childbirth, to avoid stimulation near the fetal heart.
2. Objectives:

   Primary aim:
   * To know if the application of TENS is effective in reducing pain during childbirth.

   Secondary aim:
   * To determine the most effective dose in the use of TENS in pregnant women during labor.
   * To analyze the degree of satisfaction of the pregnant women who participate in the study.
   * To evaluate whether the use of TENS reduces the dose of the painkillers during childbirth.
3. Material and Methods:

This study is a triple blind randomized trial with concealed allocation, assessor blinding for some outcomes, and intention-to-treat analysis.

It was accepted by the Ethic Committee of the Hospital Complejo Hospitalario Universitario Insular Materno Infantil of Las Palmas de Gran Canaria, Canary Islands, Spain, with registration number CEIm-CHUIMI-2016/875.

3.1. Allocation: All participants will be recruited from a group of women admitted to the hospital. If the pregnant woman meets the inclusion criteria, she will be asked to participate in the study. If yes, they must sign the informed consent, approved by the same ethical committee of the hospital.

The assignment to each group was made through the website www.random.org to perform randomization. In addition, each group has a different TENS, which has the group number. Participants in all groups will receive all the other routine obstetric care.

3.2. Sample size determination: The sample size and power calculations were performed using the software GRANMO 7.11. Calculations were based on detecting differences of 2 units in a 10 numerical pain rate scale at post-data, assuming a standard deviation of 1.9, a 2-tailed test, an alpha level of 0.05, and a desired power of 80%. These assumptions generated a sample size of 63 subjects, 21 per group.

There is a specialiced nurse that will supervised the correct functionality every day. He will be responsible for resolving dispositive problems like low charge or insufficient electrodes.

ELIGIBILITY:
Inclusion Criteria:

* Parturients with a low-risk pregnancy.
* A gestational age > 37 weeks.
* A single foetus.
* Cervical dilation of 4 cm.
* To be older than 18 years old.
* Visual deficit that causes difficulty to take the Visual Scale Analogue.

Exclusion Criteria:

* Refusal to take part in the survey.
* Failure to Sign Consent Form.
* Planned Cesarean.
* High-risk pregnancy.
* Present skin lesions in the area of the application of the electrodes.
* Pregnant with physical or mental handicap that prevents the application of the TENS device.
* Have implanted pacemakers or automatic defibrillators.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The participants will be pregnant women.
Enrollment: 63 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Pain (VAS) | - At the beginning of the use of TENS, 10 minutes later and 30 minutes later; for measuring the change of pain.
  The instrument will be used to measure the change of pain before and after the intervention will be the Visual Analogue Scale (VAS).
  Participants will be asked to mark the level of their pain on a 100 mm, no hatched VAS scale marked at one end as "no pain" and at the other as "worst pain imaginable".
Pregnant Satisfaction | Twenty-four hours postpartum, other midwife will ask participants to answer questions regarding their satisfaction with the care provided (COMFORTS scale) and if they would prefer to receive the same type of care in the future.
  The investigators will use a scale called Care in Obstetrics : measure for testing satisfaction (COMFORTS). This scale measures satisfaction during delivery and the postnatal period.
  . This scale is a valid and reliable scale to measure women's satisfaction with the care during labour and postpartum period. The investigators obtained the authorization to use the Spanish version of the COMFORTS scale.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Francisco Loro, Professor, Study Director — University of Las Palmas de Gran Canaria
Locations (1):
- University of Las Palmas de Gran Canaria, Las Palmas de Gran Canaria, Las Palmas, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lowe NK. The nature of labor pain. Am J Obstet Gynecol. 2002 May;186(5 Suppl Nature):S16-24. doi: 10.1067/mob.2002.121427. PMID 12011870
- [Background] Wong CA. Advances in labor analgesia. Int J Womens Health. 2010 Aug 9;1:139-54. doi: 10.2147/ijwh.s4553. PMID 21072284
- [Background] Simkin P, Bolding A. Update on nonpharmacologic approaches to relieve labor pain and prevent suffering. J Midwifery Womens Health. 2004 Nov-Dec;49(6):489-504. doi: 10.1016/j.jmwh.2004.07.007. PMID 15544978
- [Background] Reynolds F. Labour analgesia and the baby: good news is no news. Int J Obstet Anesth. 2011 Jan;20(1):38-50. doi: 10.1016/j.ijoa.2010.08.004. Epub 2010 Dec 13. PMID 21146977
- [Background] Lieberman E, O'donoghue C. Unintended effects of epidural analgesia during labor: a systematic review. Am J Obstet Gynecol. 2002 May;186(5 Suppl Nature):S31-68. doi: 10.1067/mob.2002.122522. PMID 12011872
- [Background] Liu EH, Sia AT. Rates of caesarean section and instrumental vaginal delivery in nulliparous women after low concentration epidural infusions or opioid analgesia: systematic review. BMJ. 2004 Jun 12;328(7453):1410. doi: 10.1136/bmj.38097.590810.7C. Epub 2004 May 28. PMID 15169744
- [Background] Anim-Somuah M, Smyth R, Howell C. Epidural versus non-epidural or no analgesia in labour. Cochrane Database Syst Rev. 2005 Oct 19;(4):CD000331. doi: 10.1002/14651858.CD000331.pub2. PMID 16235275
- [Background] Cambic CR, Wong CA. Labour analgesia and obstetric outcomes. Br J Anaesth. 2010 Dec;105 Suppl 1:i50-60. doi: 10.1093/bja/aeq311. PMID 21148655
- [Background] Jones L, Othman M, Dowswell T, Alfirevic Z, Gates S, Newburn M, Jordan S, Lavender T, Neilson JP. Pain management for women in labour: an overview of systematic reviews. Cochrane Database Syst Rev. 2012 Mar 14;2012(3):CD009234. doi: 10.1002/14651858.CD009234.pub2. PMID 22419342
- [Background] Melzack R, Wall PD. Pain mechanisms: a new theory. Science. 1965 Nov 19;150(3699):971-9. doi: 10.1126/science.150.3699.971. No abstract available. PMID 5320816
- [Background] Tournaire M, Theau-Yonneau A. Complementary and alternative approaches to pain relief during labor. Evid Based Complement Alternat Med. 2007 Dec;4(4):409-17. doi: 10.1093/ecam/nem012. PMID 18227907
- [Background] Field T. Pregnancy and labor alternative therapy research. Altern Ther Health Med. 2008 Sep-Oct;14(5):28-34. PMID 18780582
- [Background] Wang SM, Kain ZN, White P. Acupuncture analgesia: I. The scientific basis. Anesth Analg. 2008 Feb;106(2):602-10. doi: 10.1213/01.ane.0000277493.42335.7b. PMID 18227322
- [Background] Chao AS, Chao A, Wang TH, Chang YC, Peng HH, Chang SD, Chao A, Chang CJ, Lai CH, Wong AMK. Pain relief by applying transcutaneous electrical nerve stimulation (TENS) on acupuncture points during the first stage of labor: a randomized double-blind placebo-controlled trial. Pain. 2007 Feb;127(3):214-220. doi: 10.1016/j.pain.2006.08.016. Epub 2006 Oct 6. PMID 17030438
- [Background] Dowswell T, Bedwell C, Lavender T, Neilson JP. Transcutaneous electrical nerve stimulation (TENS) for pain relief in labour. Cochrane Database Syst Rev. 2009 Apr 15;(2):CD007214. doi: 10.1002/14651858.CD007214.pub2. PMID 19370680
- [Background] Santana LS, Gallo RB, Ferreira CH, Duarte G, Quintana SM, Marcolin AC. Transcutaneous electrical nerve stimulation (TENS) reduces pain and postpones the need for pharmacological analgesia during labour: a randomised trial. J Physiother. 2016 Jan;62(1):29-34. doi: 10.1016/j.jphys.2015.11.002. Epub 2015 Dec 11. PMID 26701166
- [Background] Gungor I, Beji NK. Development and psychometric testing of the scales for measuring maternal satisfaction in normal and caesarean birth. Midwifery. 2012 Jun;28(3):348-57. doi: 10.1016/j.midw.2011.03.009. Epub 2011 May 4. PMID 21546142
- [Derived] Baez-Suarez A, Martin-Castillo E, Garcia-Andujar J, Garcia-Hernandez JA, Quintana-Montesdeoca MP, Loro-Ferrer JF. Evaluation of different doses of transcutaneous nerve stimulation for pain relief during labour: a randomized controlled trial. Trials. 2018 Nov 26;19(1):652. doi: 10.1186/s13063-018-3036-2. PMID 30477529